CLINICAL TRIAL: NCT05857163
Title: Phase 3 Clinical Trial to Evaluate the Efficacy and Safety of Rifasutenizol (TNP 2198) in Combination With Rabeprazole and Amoxicillin in the Primary Treatment of Participants With H. Pylori Infection
Brief Title: Efficacy and Safety of Rifasutenizol (TNP 2198), Rabeprazole and Amoxicillin in Participants With H. Pylori Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: TenNor Therapeutics (Suzhou) Limited (Industry)
Responsible Party: Sponsor
Organization: TenNor Therapeutics Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TNP-2198-PO-07
Record Dates: First submitted 2023-04-21; First posted 2023-05-12 (Actual); Results first posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-07

CONDITIONS: H.Pylori Infection
MeSH Terms: interventions — Rabeprazole; Amoxicillin; Clarithromycin; Bismuth

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Test Group (Experimental): Rifasutenizol capsules 400 mg + Rabeprazole sodium enteric-coated tablets 20 mg + Amoxicillin capsules 1 g + Bismuth potassium citrate placebo capsules + Clarithromycin placebo tablets, twice daily (BID) for 14 days
  Interventions: Drug: Rifasutenizol capsules; Drug: Rabeprazole sodium enteric-coated tablets; Drug: Amoxicillin Capsules; Drug: Clarithromycin placebo tablets; Drug: Bismuth potassium citrate placebo capsules
- Control Group (Active Comparator): Amoxicillin capsules 1 g + Clarithromycin tablets 500 mg + Rabeprazole sodium enteric-coated tablets 20 mg + Bismuth potassium citrate capsules 240 mg + Rifasutenizol placebo capsules, BID for 14 days
  Interventions: Drug: Rabeprazole sodium enteric-coated tablets; Drug: Amoxicillin Capsules; Drug: Clarithromycin tablets; Drug: Bismuth potassium citrate capsules; Drug: Rifasutenizol placebo capsules

INTERVENTIONS:
Drug: Rifasutenizol capsules — 400 mg, BID, taken orally within half an hour after breakfast and dinner.
  Other Names: TNP-2198 capsules
  Arms: Test Group
Drug: Rabeprazole sodium enteric-coated tablets — 20 mg, BID, taken orally within half an hour before breakfast and dinner.
  Other Names: Rabeprazole
Drug: Amoxicillin Capsules — 1 g, BID, taken orally within half an hour after breakfast and dinner.
  Other Names: Amoxicillin
Drug: Clarithromycin placebo tablets — BID, taken orally within half an hour after breakfast and dinner.
  Other Names: Clarithromycin placebo
  Arms: Test Group
Drug: Bismuth potassium citrate placebo capsules — BID, taken orally within half an hour before breakfast and dinner.
  Other Names: Bismuth placebo
  Arms: Test Group
Drug: Clarithromycin tablets — 500 mg, BID, taken orally within half an hour after breakfast and dinner.
  Other Names: Clarithromycin
  Arms: Control Group
Drug: Bismuth potassium citrate capsules — 240 mg, BID, taken orally within half an hour before breakfast and dinner.
  Other Names: Bismuth
  Arms: Control Group
Drug: Rifasutenizol placebo capsules — BID, taken orally within half an hour before breakfast and dinner.
  Other Names: Rifasutenizol placebo
  Arms: Control Group

SUMMARY:
A multi-center, randomized, double-blind, bismuth-containing quadruple active comparator-controlled Phase 3 clinical study to evaluate the efficacy and safety of Rifasutenizol in combination with rabeprazole and amoxicillin in the primary treatment of participants with H. pylori infection using an adaptive design with sample size re-estimation.

DETAILED DESCRIPTION:
Subjects will be randomly assigned to test group or control group at a 1:1 ratio stratified by study site, and will receive Rifasutenizol capsules, rabeprazole sodium enteric-coated tablets, amoxicillin capsules combined with clarithromycin placebo tablets and bismuth potassium citrate placebo capsules (test group), or bismuth-containing quadruple regimen of amoxicillin capsules, clarithromycin tablets, rabeprazole sodium enteric-coated tablets and bismuth potassium citrate capsules combined with Rifasutenizol placebo capsules (control group) for 14 consecutive days.

carbon-13 (13C) UBT will be performed 4-6 weeks after the last dose to evaluate the eradication effect of H. pylori.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily sign the informed consent form.
* Age 18-65 years (inclusive), male or female.
* The result of 13C-UBT is positive (≥ 4 Delta Over Baseline), and the infection of H. pylori are confirmed by gastroscopic biopsy histology.
* Subjects agree to refrain from taking any antibiotics or traditional Chinese medicines with antibacterial effect, bismuth, and antacids (such as proton pump inhibitor, H2 receptor blocker, P-CAB) other than the study drugs during the Screening Period until the end of the study (Visit 5, i.e., Efficacy Evaluation Visit).
* Subjects and their heterosexual partners must agree to have no pregnancy plan and voluntarily take effective contraceptive measures during the trial and for at least 6 months after the end of the study medication.
* Willing to follow and able to complete all trial procedures.

Exclusion Criteria:

* Allergy to any of the study drugs (rabeprazole, amoxicillin, clarithromycin, bismuth potassium citrate), allergic constitution (multiple drug and food allergies); or any contraindication to the use of rifamycin, nitroimidazoles or study drugs.
* History of H. pylori eradication therapy (including participation in other clinical trials for H. pylori eradication).
* Subjects with confirmed tuberculosis (TB) or Mycobacterium avium complex (MAC) infection or a history of TB or MAC infection.
* History of dysphagia or any gastrointestinal disorder affecting drug absorption.
* History of obstruction pyloric; or excessive gastric acid secretion (such as Zollinger-Ellison syndrome).
* History of gastric cancer.
* History of neoplasm malignant within 5 years prior to screening, with the exception of basal cell carcinoma or carcinoma cervix in situ treated without evidence of recurrence.
* History of esophageal or gastric surgery, except for simple repair of the perforated ulcer.
* History of substance abuse or drug use within 5 years prior to screening.
* Alcohol abuse or a history of alcohol abuse within 5 years prior to screening (average weekly consumption of ≥ 14 units of alcohol: 1 unit = 285 mL of beer, or 25 mL of spirits, or 100 mL of wine/Chinese rice wine/rice wine);
* Presence of active gastric and/or duodenal ulcer.
* Anticoagulant therapy or long-term treatment with nonsteroidal anti-inflammatory drugs.
* Treatment with any other investigational new drugs within 4 weeks prior to the Screening Period.
* Any prohibited medications or non-drug therapies as specified in the protocol (see Section 10.3).
* White blood cell count or neutrophil count below the lower limit of normal range.
* Anemia (hemoglobin < 90 g/L).
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT), total bilirubin, or serum creatinine above the upper limit of normal range.
* Test positive for hepatitis B surface antigen, hepatitis C antibody, AIDS antibody, or microspironema pallidum antibody.
* Abnormal ECG with clinical significance.
* Female subjects who are pregnant, lactating, or have a positive urine pregnancy result during the Screening Period.
* Inability to communicate with the Investigator and to comply with the study requirements.
* Other conditions considered inappropriate to participate in this study by the Investigator, e.g., the subject has a history of severe central nervous system, cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal, urological, endocrine, or hematological diseases, or has clinical manifestations of these diseases.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Actual)
Dates: Start 2023-05-18 (Actual); Primary Completion 2023-12-24 (Actual); Study Completion 2024-03-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Song Z, Zhou L, Wang W, Lan C, Tang T, Xie J, Fan H, Wang X, Zuo X, Zhu Y, Liu C, Gu Y, Feng H, Gao X, Zhang Q, Zhang H, Chen J, Geng G, Ma Z; EVEREST-HP Study Group. Rifasutenizol-based triple therapy versus bismuth plus clarithromycin-based triple therapy for first-line treatment of Helicobacter pylori infection in China (EVEREST-HP): a phase 3, multicentre, randomised, triple-dummy, double-blind, controlled, non-inferiority trial. Lancet Infect Dis. 2026 Jan;26(1):101-110. doi: 10.1016/S1473-3099(25)00438-4. Epub 2025 Sep 10. PMID 40945526

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Test Group | Control Group
Started | 353 | 347
Completed | 337 | 337
Not Completed | 16 | 10

BASELINE CHARACTERISTICS:
Population: All the participants who have been randomized into groups.
Groups:
- Test Group: Rifasutenizol capsules 400 mg + Rabeprazole sodium enteric-coated tablets 20 mg + Amoxicillin capsules 1 g + Bismuth potassium citrate placebo capsules + Clarithromycin placebo tablets, BID for 14 days
- Total: Total of all reporting groups
Arm/Group | Test Group | Control Group | Total
Number analyzed (Participants) | 353 | 347 | 700
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 353 | 347 | 700
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.2 (11.68) | 39.5 (11.18) | 39.4 (11.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 220 | 219 | 439
  Male | 133 | 128 | 261
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 353 | 347 | 700
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 353 | 347 | 700
Participants with H. pylori infection [Count of Participants; unit: Participants] | 353 | 347 | 700

OUTCOME MEASURES:

1. Primary Outcome: Eradication Rate of H.Pylori Infection
Description: The eradication rate of H. pylori is defined as the percentage of participants with negative results of 13C UBT.
Time Frame: 4 to 6 weeks after the last dose of the study drugs
Population: All the participants who have been randomized into groups and received at least one dose of study drugs.
Measure: Count of Participants; unit: Participants
Arm/Group | Test Group | Control Group
Number analyzed (Participants) | 351 | 346
Participants | 323 | 304

2. Secondary Outcome: Eradication Rate of Antibiotic-resistant Strains of H.Pylori
Description: Percentage of Participants with Successful Helicobacter Pylori (H.pylori) Eradication in Participants with antibiotic-resistant Strains of H.pylori at Baseline (based on the test results of 13C UBT)
Time Frame: 4 to 6 weeks after the last dose of the study drugs
Population: Participants who have been randomized into groups and received at least one dose of study drugs.
Measure: Count of Participants; unit: Participants
Arm/Group | Test Group | Control Group
Number analyzed (Participants) | 351 | 346
Participants
  Clarithromycin resistant: number analyzed (Participants) | 107 | 129
  Clarithromycin resistant | 92 | 105
  Clarithromycin susceptible: number analyzed (Participants) | 179 | 164
  Clarithromycin susceptible | 169 | 154
  Metronidazole resistant: number analyzed (Participants) | 186 | 209
  Metronidazole resistant | 168 | 182
  Metronidazole susceptible: number analyzed (Participants) | 99 | 84
  Metronidazole susceptible | 92 | 77
  Amoxicillin resistant: number analyzed (Participants) | 20 | 27
  Amoxicillin resistant | 19 | 24
  Amoxicillin susceptible: number analyzed (Participants) | 266 | 266
  Amoxicillin susceptible | 242 | 235
  Levofloxacin resistant: number analyzed (Participants) | 101 | 102
  Levofloxacin resistant | 93 | 85
  Levofloxacin susceptible: number analyzed (Participants) | 184 | 191
  Levofloxacin susceptible | 167 | 174
  Clarithromycin & Amoxicillin resistant: number analyzed (Participants) | 13 | 18
  Clarithromycin & Amoxicillin resistant | 12 | 16
  DR (drug-resistant) defined as resistant to at least one class antibiotics for H. pylori infection: number analyzed (Participants) | 243 | 250
  DR (drug-resistant) defined as resistant to at least one class antibiotics for H. pylori infection | 221 | 218
  MDR (multidrug-resistant) resistant to at least two classes of antibiotics for H. pylori infection: number analyzed (Participants) | 119 | 149
  MDR (multidrug-resistant) resistant to at least two classes of antibiotics for H. pylori infection | 107 | 121

3. Secondary Outcome: Safety by Assessment of the Number of Participants With Adverse Events (AEs)
Description: An Adverse Event (AE) is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An Adverse Event can therefore be any unfavorable and unintended sign (including abnormal laboratory values or abnormal clinical test results), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as Adverse Events.
Time Frame: up to 4-6 weeks after the last dose of the study drugs
Population: All the participants who have been randomized into groups and received at least one dose of study drugs.
Measure: Count of Participants; unit: Participants
Arm/Group | Test Group | Control Group
Number analyzed (Participants) | 351 | 346
Participants | 131 | 184

4. Secondary Outcome: Time to Reach the Maximum Observed Plasma Concentration (Tmax) of Rifasutenizol (TNP-2198) on Day 1
Description: Plasma concentrations of Rifasutenizol (TNP-2198) were measured by a specific and validated assay. Plasma pharmacokinetic (PK) parameters of Rifasutenizol (TNP-2198) were read directly from the plasma concentration versus time profiles or calculated by using standard non-compartmental methods.
Time Frame: Day 1: 30 minutes before and 1, 2, 3, 4, 5, 6, 7, 8, 10, and 12 hours after Rifasutenizol (TNP-2198) administration
Population: All randomized participants who have received Rifasutenizol (TNP-2198) and have at least one pharmacokinetic parameter data.
Measure: Median (Full Range); unit: h
Arm/Group | Test Group
Number analyzed (Participants) | 20
h | 4.08 [1.00 to 5.08]

5. Secondary Outcome: Time to Reach the Maximum Observed Plasma Concentration (Tmax) of Rifasutenizol (TNP-2198) on Day 14
Description: Plasma concentrations of Rifasutenizol (TNP-2198) were measured by a specific and validated assay. Plasma PK parameters of Rifasutenizol (TNP-2198) were read directly from the plasma concentration versus time profiles or calculated by using standard non-compartmental methods.
Time Frame: Day 14: 30 minutes before and 1, 2, 3, 4, 5, 6, 7, 8, 10, 12 hours after Rifasutenizol (TNP-2198) administration
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: h
Arm/Group | Test Group
Number analyzed (Participants) | 20
h | 4.58 [1.00 to 5.08]

6. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Rifasutenizol (TNP-2198) on Day 1
Description: as for outcome 5
Time Frame: Day 1: 30 minutes before and 1, 2, 3, 4, 5, 6, 7, 8, 10, 12 hours after Rifasutenizol (TNP-2198) administration
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Test Group
Number analyzed (Participants) | 20
ng/mL | 324 (145)

7. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Rifasutenizol (TNP-2198) on Day 14
Description: as for outcome 5
Time Frame: Day 14: 30 minutes before and 1, 2, 3, 4, 5, 6, 7, 8, 10, 12 hours after Rifasutenizol (TNP-2198) administration
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Test Group
Number analyzed (Participants) | 20
ng/mL | 504 (187)

8. Secondary Outcome: Half Life (t1/2) of Rifasutenizol (TNP-2198) on Day 1
Description: as for outcome 5
Time Frame: Day 1: 30 minutes before and 1, 2, 3, 4, 5, 6, 7, 8, 10, 12 hours after Rifasutenizol (TNP-2198) administration
Population: as for outcome 4
Measure: Median (Full Range); unit: h
Arm/Group | Test Group
Number analyzed (Participants) | 20
h | 3.25 [2.21 to 5.25]

9. Secondary Outcome: Half Life (t1/2) of Rifasutenizol (TNP-2198) on Day 14
Description: as for outcome 5
Time Frame: Day 14: 30 minutes before and 1, 2, 3, 4, 5, 6, 7, 8, 10, 12 hours after Rifasutenizol (TNP-2198) administration
Population: as for outcome 4
Measure: Median (Full Range); unit: h
Arm/Group | Test Group
Number analyzed (Participants) | 20
h | 3.05 [2.45 to 5.80]

10. Secondary Outcome: Area Under the Plasma Concentration-time Curve Within a Dosing Interval (AUC0-tau) of Rifasutenizol (TNP-2198) on Day 1
Description: as for outcome 5
Time Frame: Day 1: 30 minutes before and 1, 2, 3, 4, 5, 6, 7, 8, 10, 12 hours after Rifasutenizol (TNP-2198) administration
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Test Group
Number analyzed (Participants) | 20
h*ng/mL | 1160 (507)

11. Secondary Outcome: Area Under the Plasma Concentration-time Curve Within a Dosing Interval (AUC0-tau) of Rifasutenizol (TNP-2198) on Day 14
Description: as for outcome 5
Time Frame: Day 14: 30 minutes before and 1, 2, 3, 4, 5, 6, 7, 8, 10, 12 hours after Rifasutenizol (TNP-2198) administration
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Test Group
Number analyzed (Participants) | 20
h*ng/mL | 1950 (737)

12. Secondary Outcome: Area Under the Plasma Concentration-time Curve From the Time of Administration Extrapolated to Infinity (AUC0-∞) of Rifasutenizol (TNP-2198) on Day 1
Description: as for outcome 5
Time Frame: Day 1: 30 minutes before and 1, 2, 3, 4, 5, 6, 7, 8, 10, 12 hours after Rifasutenizol (TNP-2198) administration
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Test Group
Number analyzed (Participants) | 20
h*ng/mL | 1240 (548)

13. Secondary Outcome: Area Under the Plasma Concentration-time Curve From the Time of Administration Extrapolated to Infinity (AUC0-∞) of Rifasutenizol (TNP-2198) on Day 14
Description: as for outcome 5
Time Frame: Day 14: 30 minutes before and 1, 2, 3, 4, 5, 6, 7, 8, 10, 12 hours after Rifasutenizol (TNP-2198) administration
Population: All randomized participants who have received Rifasutenizol (TNP-2198) and have at least one pharmacokinetic
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Test Group
Number analyzed (Participants) | 20
h*ng/mL | 2160 (819)

14. Secondary Outcome: Volume of Distribution (Vd/F) of Rifasutenizol (TNP-2198) on Day 1
Description: as for outcome 5
Time Frame: Day 1: 30 minutes before and 1, 2, 3, 4, 5, 6, 7, 8, 10, 12 hours after Rifasutenizol (TNP-2198) administration
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Test Group
Number analyzed (Participants) | 20
mL | 2010000 (1200000)

15. Secondary Outcome: Volume of Distribution (Vd/F) of Rifasutenizol (TNP-2198) on Day 14
Description: as for outcome 5
Time Frame: Day 14: 30 minutes before and 1, 2, 3, 4, 5, 6, 7, 8, 10, 12 hours after Rifasutenizol (TNP-2198) administration
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Test Group
Number analyzed (Participants) | 20
mL | 1310000 (982000)

16. Secondary Outcome: Clearance (CL/F) of Rifasutenizol (TNP-2198) on Day 1
Description: as for outcome 5
Time Frame: Day 1: 30 minutes before and 1, 2, 3, 4, 5, 6, 7, 8, 10, 12 hours after Rifasutenizol (TNP-2198) administration
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mL/h
Arm/Group | Test Group
Number analyzed (Participants) | 20
mL/h | 425000 (298000)

17. Secondary Outcome: Clearance (CL/F) of Rifasutenizol (TNP-2198) on Day 14
Description: as for outcome 5
Time Frame: Day 14: 30 minutes before and 1, 2, 3, 4, 5, 6, 7, 8, 10, 12 hours after Rifasutenizol (TNP-2198) administration
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mL/h
Arm/Group | Test Group
Number analyzed (Participants) | 20
mL/h | 252000 (172000)

ADVERSE EVENTS:
Time Frame: up to 4-6 weeks after the last dose of the study drugs
Arm/Group | Test Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/351 | 0/346
Serious Adverse Events (participants affected / at risk) | 2/351 | 2/346
Other Adverse Events (participants affected / at risk) | 65/351 | 143/346
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Test Group (N=351) | Control Group (N=346)
Vertigo positional (Ear and labyrinth disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Sclerosing pneumocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0
Defaecation disorder (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Test Group (N=351) | Control Group (N=346)
Diarrhoea (Gastrointestinal disorders) | 24 | 19
Nausea (Gastrointestinal disorders) | 22 | 21
Dizziness (Nervous system disorders) | 21 | 12
Dysgeusia (Nervous system disorders) | 17 | 125

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-14): https://cdn.clinicaltrials.gov/large-docs/63/NCT05857163/Prot_SAP_000.pdf